CLINICAL TRIAL: NCT01051011
Title: A Multi-center, Randomized, Open-label, Active-controlled Study to Compare the Safety, Tolerability and Effect on Glycemic Control of Taspoglutide Versus Insulin Glargine in Insulin-naive Type 2 Diabetic Patients Inadequately Controlled With Metformin and Sulphonylurea Combination Therapy.
Brief Title: A Study to Compare Taspoglutide and Insulin Glargine in Insulin-Naïve Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin and Sulfonylurea Combination Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: high discontinuation rates mainly due to GI tolerability and implementation of risk mitigation plan to address hypersensitivity reactions
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZC22565
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin; taspoglutide

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: metformin; Drug: taspoglutide
- 2 (Experimental)
  Interventions: Drug: metformin; Drug: taspoglutide
- 3 (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: metformin

INTERVENTIONS:
Drug: insulin glargine — initial dose 10 international units (IU) sc daily, titrated according to the mean FPG, 24 (-52) weeks
  Arms: 3
Drug: metformin — as prescribed
Drug: taspoglutide — 10mg sc weekly, 24 (-52) weeks
  Arms: 1
Drug: taspoglutide — 10mg sc weekly the 1st 4 weeks followed by 20mg sc weekly, 24 (-52) weeks
  Arms: 2

SUMMARY:
This randomized, open-label, parallel arm study will compare the safety, tolerability and effect on glycemic control of taspoglutide versus insulin glargine in insulin-naïve patients with type 2 diabetes mellitus inadequately controlled on merformin and sulfonylurea combination therapy. Patients will be randomized to receive either taspoglutide 10mg subcutaneously (sc) weekly, or taspoglutide 10mg sc weekly for 4 weeks followed by 20mg sc weekly, or insulin glargine at an initial dose of 10 international units sc daily. Metformin treatment will be continued in all patients throughout the study, whereas sulfonylurea will be discontinued before starting study treatment. Anticipated time on study treatment is 24 weeks, with an option to continue the assigned treatment for another 28 weeks. Target sample size is 500-600 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age
* type 2 diabetes mellitus, treated with stable dose of metformin and sulfonylurea for >/= 12 weeks prior to screening
* HbA1c 7-10% at screening
* body weight stable (+/-5%) for >/= 12 weeks prior to screening
* fasting C-peptide >/=1ng/ml
* treatment-naïve for insulin

Exclusion Criteria:

* diagnosis or history of type 1 diabetes mellitus or secondary forms of diabetes
* acute metabolic diabetic complications or evidence of clinically significant diabetic complications
* clinically symptomatic gastrointestinal disease
* history of chronic pancreatitis or acute idiopathic pancreatitis
* >3 episodes of severe hypoglycemia within 6 months prior to screening
* miocardial infarcion, unstable angina pectoris, coronary artery bypass surgery, post-transplantation cardiomyopathy or stroke within 6 months prior to screening
* any treatment with exenatide, exendin analogues, GLP-1 or its analogues

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Glycemic control assessed by HbA1c | week 24

SECONDARY OUTCOMES:
Fasting plasma glucose, incidence of hypoglycemia, proportion of patients achieving target HbA1c | week 24
Body weight, lipid profile (triglycerides, total cholesterol, LDL and HDL cholesterol, LDL/HDL ratio) | week 24
Safety and tolerability: Adverse events (including hypoglycemia), vital signs, laboratory parameters | throughout study, laboratory assessments weeks 12, 24, 32 and 52
Meal tolerance test (in a subset of patients): Glucose, insulin, C-peptide, glucagon values | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- China (13):
  - Beijing
  - Beijng
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Hefei
  - Nanjing
  - Nanning
  - Shanghai
  - Shijiazhuang
  - Tianjin
  - Tianjin (天津)
- Hong Kong, Hong Kong
- Malaysia (6):
  - George Town
  - Johor Bahru
  - Kelantan
  - Kuala Lumpur
  - Kuala Selangor
  - Putrajaya
- Philippines (4):
  - Cebu
  - Iloilo City
  - Manila
  - Pasig
- South Korea (7):
  - Busan
  - Daegu
  - Gyeonggi-do
  - Incheon
  - Kangwon-do
  - Kyounggi-do
  - Seoul
- Taiwan (5):
  - Chia-Yi City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Nakhonratchasima